CLINICAL TRIAL: NCT03228303
Title: Nilotinib Versus Imatinib in Treatment of Patients With Newly Diagnosed Chronic Myeloid Leukemia
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Jean George Maxwell, ClinIcal professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Jgmaxwell
Record Dates: First submitted 2017-07-16; First posted 2017-07-24 (Actual); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib; Imatinib Mesylate

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chronic phase CML treated by nilotinib (Active Comparator): Newly diagnosed
  Interventions: Drug: Nilotinib 150 MG [Tasigna]
- Chronic phase CML treated by imatinib (Active Comparator): Newly diagnosed
  Interventions: Drug: Imatinib 400mg

INTERVENTIONS:
Drug: Nilotinib 150 MG [Tasigna] — Nilotinib vs imatinib in patients with newly diagnosed CML-CP
  Arms: Chronic phase CML treated by nilotinib
Drug: Imatinib 400mg — Nilotinib vs imatinib in patients with newly diagnosed CML-CP
  Arms: Chronic phase CML treated by imatinib

SUMMARY:
Nilotinib vs imatinib in patients with newly diagnosed CML-CP

DETAILED DESCRIPTION:
Study size is 100 patients in 2 arms 50 patients in nilotinib ttt 50 patients in imatinib ttt

ELIGIBILITY:
Inclusion Criteria:

* chronic phase CML not received treatment
* Pts with no heart disease
* Pts with no abnormal cholesterol level

Exclusion Criteria:

* Any pts treated before with diff. Treatment
* Pts. With past history of heart problems
* Pts. With abnormal cholesterol level

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Nilotinib vs imatinib in patients with newly diagnosed CML-CP: Overall survival rate in years | 3 years cutoff
  Overall survival rate in years
Nilotinib vs imatinib in patients with newly diagnosed CML-CP: Cholesterol level in mg | 3 years cutoff
  cholesterol level in mg
Nilotinib vs imatinib in patients with newly diagnosed CML-CP: Heart state by assessment by ECG | 3 years cutoff
  heart state by assessment by ECG
Nilotinib vs imatinib in patients with newly diagnosed CML-CP: Free survival rate in years | 3 years cutoff
  free survival rate in years